CLINICAL TRIAL: NCT04494139
Title: Acceptability, Feasibility and Effectiveness of a Worksite Intervention to Lower Cardiometabolic Risk in South Africa
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Durban University of Technology (Other)
Collaborators: Yale University (Other); Dhulikhel Hospital (Other)
Responsible Party: Principal Investigator, Dr Ashika Naicker, Senior Lecturer, Durban University of Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IREC173/18
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Dietary Intervention; Pre Diabetes; Hypertension
Keywords: Pre diabetes; Canteen intervention; Behavioral intervention
MeSH Terms: conditions — Glucose Intolerance; Hypertension

STUDY DESIGN:
Intervention Model Description: Arm 1: Canteen only intervention Arm 2: Canteen and behavioral intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Canteen Only (Active Comparator): Train canteen staff and implement canteen intervention in the canteen space: interventions targeting food quality and quantity, intervention targeting food choice at point of sale, interventions target improved supply, interventions targeting price and promotional material.
  Interventions: Other: Canteen
- Behavioral and Canteen intervention (Experimental): The behavioral intervention will be comprised of a combination of intensive education sessions and goal setting and monitoring based on a validated worksite curriculum tailored to local needs. The curriculum includes 24 sessions: 16 core weekly sessions during the first four months of the intervention followed by 8 weekly maintenance sessions (text messages). Each session will be facilitated by a nutritionist/dietitian and a peer educator; and will last one hour. Broadly, the curriculum covers the subject matters of importance of healthy weight, eating a healthy diet, increasing physical activity, stress management, and challenges of lifestyle changes. Participants will be encouraged to keep food and activity diaries throughout the course of the study. During the maintenance period, the focus will be on overcoming declines in motivation and on maintaining long-term healthy behaviors.
  Interventions: Behavioral: Behavioral and Canteen intervention; Other: Canteen

INTERVENTIONS:
Behavioral: Behavioral and Canteen intervention — Behavioral intervention: 16 weeks
  Arms: Behavioral and Canteen intervention
Other: Canteen — Canteen changes to introduce health foods

SUMMARY:
As an important way to translate cardiovascular disease prevention efforts, worksite interventions can facilitate healthy food choices, health education, and social support. This proposed project is adapted and scaled-up from the Nepal study, and will measure the effectiveness of a canteen and a behavioral intervention on cardio-metabolic risk at a worksite in South Africa. This study will estimate the added benefit of a proven individual-level dietary intervention over environmental-level changes for preventing cardio-metabolic risk within the South African context. If the study demonstrates a significant effect, a scaled-up approach could produce an important reduction in cardiovascular disease burden through environmental and individual level prevention programs in South Africa.

DETAILED DESCRIPTION:
The effectiveness of the multi-component environmental worksite intervention will be measured by evaluating the change in number of individuals attaining two or more cardiometabolic risk reduction goals (i.e., reductions in HbA1c, blood pressure, triglycerides, cholesterol and weight). Secondary outcomes will include the individual changes in the risk factors included in the primary outcome, as well as in cardiometabolic risk not included in the composite score (i.e., LDL, HDL, total cholesterol/HLD ratio), in dietary intake, in physical activity, and in worksite-level food and beverage sales.

Specific objectives is as follows:

1. To measure the effectiveness of a canteen intervention on a composite score based upon improvement in cardio-metabolic risk factors (0-3) with success defined by HbA1c decrease ≥0.5%; a systolic blood pressure decrease ≥5 mmHg; and a decrease in plasma triglycerides ≥10 mg/dl. We will compare the change in the score after six months of the canteen intervention to the baseline results.
2. To measure the effectiveness of a behavioral intervention on a composite score based upon improvement in cardio-metabolic risk factors (0-3) with success defined by HbA1c decrease ≥0.5%; a systolic blood pressure decrease ≥5 mm Hg. We will compare the change in the score in behavior intervention group to the baseline results.
3. To measure the effectiveness of a canteen intervention on diabetes risk (By comparing the change in HbA1c of participants after six months of canteen intervention to the baseline results).
4. To measure the effectiveness of a behavioral intervention on diabetes risk (By comparing the change in HbA1c of participants after six months of behavior plus canteen intervention to the change over six months during the canteen only intervention).
5. To measure the combined effect of canteen and behavioral intervention on diabetes risk (By comparing the change in HbA1c levels of the participants of canteen plus behavioral intervention to baseline results).
6. To measure the effectiveness of a canteen intervention on dietary behavior (By comparing change in the proportion of healthy foods adopted by the participants after six months of canteen intervention to the change in the proportion of healthy food consumption at baseline).
7. To measure the effectiveness of a behavioral intervention on dietary behavior (By comparing the change in the proportion of healthy foods eaten by the participants after six months of behavior plus canteen intervention to the change over six months during the canteen only intervention) Interventions The study will recruit 350 employees at a worksite in Durban, Kwa Zulu Natal using the worksite characteristic checklist for best fit to the study. Formative work will be done to determine the best fit for the implementation of the intervention to the worksite. At baseline, 6 months, 12 months and 18 months, standard questionnaire will be administered to record relevant characteristics of the participants, physical activity, smoking, stress, alcohol intake and diet. Food sales data will be abstracted from the administrative database of the canteen. Blood samples will be collected and analyzed for HbA1c, fasting glucose, and lipid profile (HDL, LDL, total cholesterol, triglycerides). Participants height, weight, waist circumference, hip circumference, and blood pressure will be measured. After 6 months of control period, the participants will receive the canteen intervention. After six months of the canteen/physical environment intervention, half of the participants will be randomized to receive a canteen and behavioral intervention; whereas the other half receives canteen only intervention. The behavioral intervention will be comprised of a combination of intensive education sessions and goal setting and monitoring based on a validated worksite curriculum tailored to local needs. The curriculum will include 24 sessions: 16 core weekly sessions during the first four months of the intervention followed by 8 weekly maintenance sessions (text messages). Each session will be facilitated by a nutritionist/dietitian and a peer educator; and will last one hour. Broadly, the curriculum will cover the subject matters of importance of healthy weight, eating a healthy diet, increasing physical activity, stress management, and challenges of lifestyle changes. Participants will be encouraged to keep food and activity diaries throughout the course of the study. During the maintenance period, the focus will be on overcoming declines in motivation and on maintaining long-term healthy behaviors. Participants will set at least two lifestyle change goals such as consuming half of the total grains as whole grains, walking 30 minutes a day, reducing 7% of the body weight, and similar goals to achieve during the sessions based on their baseline CVD profile. Participants will be followed up at 6 months (at the end of step 1 intervention), 12 months (at the end of step 2 intervention). During each follow up, fasting blood samples will be collected and analyzed for HbA1c, fasting glucose, and lipid profile (HDL, LDL, total cholesterol, triglycerides).

The primary analysis will use chi squared test use to compare (a) Proportion of individual with score ≥ 2 during canteen only intervention to the proportion of individual with score ≥ 2 during the control period; (b) Proportion of individual with score ≥ 2 during canteen and behavioral intervention to the proportion of individual with score ≥ 2 during canteen only intervention. Logistic regression for the proportion of individual with score ≥ 2 as outcome and canteen only vs canteen and behavioural as exposure will be conducted. Secondary analysis will use paired t-test to compare (a) the change in healthy food intake and HbA1c during canteen only intervention to the change in healthy food intake and HbA1C during the control period (b) the change in healthy food intake and HbA1C% during canteen and behavioral intervention to the change in healthy food intake and HbA1C% during canteen only intervention.

The following process outcomes will be measured:

1. Program adoption will be measured by quantifying workers participation through calculating the percentages of total employees agreeing to screening, and percentages agreeing to participate in the intervention.
2. Program fidelity will be determined by measuring changes in the worksite environment, and management support for the program. To assess compliance to the recommended dietary interventions (i.e., provide healthy food options in the canteen, eliminate SSBs) every month in the intervention period, a member of the study team not affiliated with the worksite will do a random audit.
3. Program feasibility will be measured by quantifying the changes in sales of healthy and unhealthy foods and beverages at the canteen from baseline to follow-up.
4. Program adoption and acceptability will be assessed through focus group discussions with employees (lifestyle participants and lifestyle drop outs) managers and non-eligible participants on worksite environmental changes.
5. The value and return on investment of the intervention for employers will be measured by assessing program cost and cost-effectiveness and changes in staff productivity, absenteeism, health status, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Full time employees
* 18 years or above of age
* No confirmation of diabetes and, not on diabetes medication OR Have HbA1c of 5.7% to 6.4%. OR Prediabetes group with FBS of 100- 126 mg/dL Systolic blood pressure 120 mm Hg or more or Diastolic blood pressure 80 mm Hg or more and not on blood pressure medication

Exclusion Criteria:

* Less than 18 years
* On diabetes medication
* On hypertension medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Cardiometabolic Risks | six months
  A composite score based upon improvement in 3 cardio-metabolic risk factors (0-3) [HbA1c decrease ≥0.5%; a systolic blood pressure decrease (SBP) ≥5 mm Hg; and plasma triglycerides decrease ≥10 mg/d
Healthy food intake | Six months
  Intake of whole grains, fruits and vegetables and other healthy labelled items in the canteen from sales data

SECONDARY OUTCOMES:
Hba1c | Six months
  Glycated haemoglobin, % continuous variable
Systolic Blood pressure | Six months
  An average of three measurements, mmHg continuous variabl

CONTACTS AND LOCATIONS:
Overall Officials: Ashika Naicker, PhD, Principal Investigator — Durban University of Technology

IPD SHARING:
Plan to Share IPD: No